CLINICAL TRIAL: NCT05973201
Title: Evaluation De La Réalité Virtuelle Pour Réduire L'anxiété, La Douleur Et De La Durée D'une Fibroscopie Bronchique Vigile Non Urgente En Soins Critiques
Brief Title: Evaluation of Virtual Reality to Reduce Anxiety, Pain and Duration of Non-emergency Vigile Bronchial Fibroscopy (AVATAR)
Acronym: AVATAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP220834; PHRIP-21-0055 (Other Grant/Funding Number: French ministry of health); 2023-A00163-42 (Other: IDRCB)
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Disorder; Lung Infection
Keywords: Virtual reality; Pulmonary fibroscopy; Anxiety; Pain; Intensive care
MeSH Terms: conditions — Respiration Disorders; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Patients in whom elective BF has been scheduled and who have given consent to the study will be randomised (1:1) to either the control group (BF after local anaesthesia (LA)) or the experimental group (BF after AL and VR immersion). Randomization will be done 30 minutes before BF, after an initial assessment of anxiety (pre-BF VAS) and will be stratified according to whether or not a psychotropic drug and/or a level II analgesic is taken the day before or on the day of BF.
  The randomization list will be programmed in advance by the study statistician using SAS software and will be generated and edited by another statistician independent of the study from the HEGP clinical research unit. The randomization list will be kept by the study sponsor (AP-HP). It will be available to users via web-based software (CleanWeb software (Telemedicine Technologies, http: //www.tentelemed.com/la-solution-cleanweb/)].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional arm (Experimental): Fibroscopy performed under local anesthesia with immersion in a virtual reality scenario
  Interventions: Device: Virtual reality headset
- Conventional arm (No Intervention): Fibroscopy performed under local anesthesia without immersion in a virtual reality scenario

INTERVENTIONS:
Device: Virtual reality headset — A HEALTHY MIND® brand VR headset is dedicated to the study. The kit includes a noise-reducing audio headset, a face mask diffusing the visual part, a touchscreen tablet connected to the two VR headset systems, and a microphone connected to the tablet.
  The available software allows patients to choose between 5 natural environments in which a hypnotic speech is broadcast, available in several languages (French, English, Spanish, Russian, Arabic).
  Arms: interventional arm

SUMMARY:
Bronchial fibroscopy (BF) is a routine practice examination in critical care areas. It can be useful either for the diagnosis of the causal pathology of respiratory distress or for the diagnosis of lung infection, sometimes nosocomial. In patients in spontaneous and conscious ventilation, BF are performed vigil after local anesthesia according to the recommendations of the Société de Pneumologie de langue Française. The good tolerance of the examination and its good conduct may require the use of anxiolytics, sedatives or analgesics to limit the traumatic experience of a highly anxiety-provoking examination. Virtual reality (VR) combines a set of paramedical techniques (hypnosis, music therapy, sophrology) and is now a non-drug alternative to improve the tolerance of certain invasive gestures.VR has been shown to reduce pain and anxiety during first pathways placement or digestive endoscopies. To date, there is no evidence of the benefit of VR when performing semi-urgent BF in critical care areas.

DETAILED DESCRIPTION:
Bronchial fibroscopy (BF) is an invasive examination mainly performed in vigilant patients under local anesthesia very regularly performed in patients hospitalized in critical care. Despite local anesthesia, and paradoxically also because of local anesthesia that makes the airflow in the upper airway imperceptible, BF is an anxiety-provoking and sometimes uncomfortable examination. Drug options are offered by physicians on a case-by-case basis and in response to patients' discomfort or anxiety. We believe that a preventive, non-drug strategy would improve comfort, reduce anxiety and improve patients' experience during BF. To reduce anxiety and improve patient comfort, there are non-drug alternatives such as hypnosis, music therapy or virtual reality. Hypnosis requires the availability of previously trained caregivers and a calm environment. Music therapy is difficult to apply in IS because of pre-existing noise pollution. We hypothesize that virtual reality would reduce patient anxiety during a bronchial fibroscopy in bed in critical care, improve the patient and caregiver experience and optimize its realization. Virtual reality (VR) is a technology that allows the patient to be projected, via a computer system, into an immersive virtual world. The patient's immersion in the virtual environment is accompanied by the feeling of "presence" which can be defined as the authentic feeling of existing in a world other than the one where the body is physically located.This specificity, coupled with the ability to isolate the patient's visual and auditory field, make this tool a promising solution to improve the well-being of patients during the care offer. VR is distributed by a set of devices to digitally simulate an environment mobilizing the different senses of its user: sight most often but possibly also touch, hearing or smell. VR, most often distributed via video and audio headset, is a complete immersive experience that can bring together hypnotic scenario and music therapy.

HEALTHY MIND® has designed a VR headset to relieve pain and anxiety in patients in healthcare facilities in a non-drug way. Indeed, this helmet has been developed to exercise analgesic and anxiolytic actions through specific virtual environments by combining different principles such as medical hypnosis, music therapy, light therapy and cardiac coherence. The proposed immersion themes combined with breathing exercises in the initial phase, generate better stress management.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years of age)
* Hospitalized in a critical care unit (intensive care and intensive care)
* Conscious (Glasgow score >13)
* Spontaneous ventilation
* Requiring the realization of a FB
* First BF during hospitalization
* Having signed a consent to participate in the study
* Affiliation to social security

Exclusion Criteria:

* Non-French-speaking patient
* Protected minors or adults who cannot consent to participate
* People with major neurocognitive impairment
* Patient refusing to participate in the study
* Patient on State medical aid
* Patient under guardianship or curatorship or under judicial protection
* BF for a vital emergency
* Prior inclusion in the study
* Pregnant or breastfeeding women
* Presence of a tracheostomy or tracheostomy
* Participation in other intervention research
* Epilepsy
* Visual impairment (blindness) or severe hearing impairment (hearing loss, deafness) that does not allow the use of the helmet
* Psychiatric pathologies such as delusional disorders, hallucinations or schizophrenia.
* Autism spectrum disorders
* Patient sensitive to motion sickness
* Refractory migraine under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Maximum value of patient's anxiety experienced during BF assessed by the visual analogue scale (VAS) immediately after the BF | Immediately after BF
  The visual analogue scale is a rating scale in the form of a 10 cm strip graduated in mm that can be presented horizontally or vertically. On the face presented to the patient, there is a cursor that he mobilizes on a straight line with one end corresponding to "absence of anxiety" and the other to "maximum anxiety imaginable". The patient must then place the cursor where he locates his anxiety. VAS ranges from 0 to 100 mm.

SECONDARY OUTCOMES:
The relative change of patient's anxiety before and after BF assessed by the STAI-A scale (state anxiety scale) | Immediately after BF
  The Spielberger State-Trait Anxiety Inventory (STAI) is a 40-item self-report measure of anxiety using a 4-point Likert-type scale (from 1 to 4 points) for each item. It has two scales: State anxiety, i.e. how one feels at the moment; and Trait anxiety, i.e. how one generally feels. Both scales consist of 20 items. The state scale has 10 reverse-scored items, the trait scale has 7. Scores of both scales ranges from 20 to 80.
Patient's anxiety when leaving the intensive care unit (or on the 7th day at the latest, after BF) assessed by the visual analogue scale (VAS) | When leaving the intensive care unit or on the 7th day at the latest, post BF
  The visual analogue scale is a rating scale in the form of a 10 cm strip graduated in mm that can be presented horizontally or vertically. On the face presented to the patient, there is a cursor that he mobilizes on a straight line with one end corresponding to "absence of anxiety" and the other to "maximum anxiety imaginable". The patient must then place the cursor where he locates his anxiety. VAS ranges from 0 to 100 mm.
Maximum value of patient's pain experienced during BF assessed by the visual analogue scale (VAS) immediately after the FB | Immediately after BF
  The visual analogue scale is a rating scale in the form of a 10 cm strip graduated in mm that can be presented horizontally or vertically. On the face presented to the patient, there is a cursor that he mobilizes on a straight line with one end corresponding to "absence of pain" and the other to "maximum pain imaginable". The patient must then place the cursor where he locates his pain. VAS ranges from 0 to 100 mm.
Patient's pain experienced during BF evaluated by the nursing staff assessed by the ALGOPLUS scale immediately after the FB | Immediately after BF
  The ALGOPLUS scale was specifically developed to evaluate and manage acute pain in the elderly in all situations in which reliable self-assessment is not feasible. The scale is composed of 5 items (observational areas/domains). Each item checked "yes" is accorded 1 point and the sum of checked items gives a total score ranging from 1 to 5.
The relative change of patient's maximum pulse measured during BF compared to pulse measured before BF | Immediately after BF
  The relative change of patient's maximum pulse measured during BF compared to pulse measured before BF
The relative change of patient's maximum respiratory rate measured during BF compared to respiratory rate measured before BF | Immediately after BF
  The relative change of patient's maximum respiratory rate measured during BF compared to respiratory rate measured before BF
The relative change of patient's maximum blood pressure measured during BF compared to blood pressure measured before BF | Immediately after BF
  The relative change of patient's maximum blood pressure measured during BF compared to blood pressure measured before BF
The duration of BF (in minutes) from the start of the local anesthesia to the permanent removal of the fibroscopy | Immediately after BF
  The duration of BF (in minutes) from the start of the local anesthesia to the permanent removal of the fibroscopy
Tolerance to the VR assessed by a questionnaire measuring the side effects of the VR | 1 day post BF
  The questionnaire items lists the side effects of the VR (8 items with 3 answer categories: yes, no and do not know).
Patient anxiety experienced before BF evaluated by the nursing staff assessed by Hamilton scale | Before BF
  The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety.The scale consists of 14 items designed to assess the severity of a patient's anxiety.
The total dose of sedative and anxiolytic drugs administered during BF | Immediately after BF
  The total dose of midazolam, alprazolam, hydroxyzine, diprivan, stage II or III analgesics administered during BF
The quality of FB (specific questionnaire completed by the physician describing the quality of exploration, the possibility of taking samples and the satisfaction VAS). | Immediately after BF
  A specific questionnaire completed by the physician in charge of the BF will be used describing the quality of the exploration and the possibility of taking samples
Remote patient satisfaction with FB measured using the e-SATIS ?questionnaire (Haute Autorité de Santé "prise en charge" section), and the answer to the single question: "Would you have a bronchial fibroscopy again in the future) | 7 days post BF
  E-SATIS is an experience and satisfaction questionnaire, in which all patients are invited to participate, following treatment in a health establishment, hospital or clinic. The questionnaire is validated by the French Haute autorité de santé. The "patient care" section of the questionnaire was used to assess remote patient's satisfaction on the BF procedure. For each responding patient, a score ranging from 1 [bad experience] to 5 [excellent experience] (transformed into a value from 0 to 100) is given to each of his answers.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra GOMES, Nurse, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - CHI Aix en Provence, Aix-en-Provence
  - CHU Dijon, Dijon
  - Hôpital Le Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital européen Georges Pompidou - AP-HP, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR)